CLINICAL TRIAL: NCT04882995
Title: Effect of Preoperative Fiber on Postoperative Bowel Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Deepali Maheshwari, Clinical Instructor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H00017494
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Constipation; Prolapse, Vaginal
Keywords: Postoperative constipation
MeSH Terms: conditions — Constipation; Uterine Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - Received fiber (Experimental): Participants received 14 doses of psyllium fiber packet (Metamucil, 3.4g). They were instructed to take 1 packet twice a day beginning 7 days before surgery.
  Interventions: Dietary Supplement: Psyillium fiber
- Control - Did not receive fiber (No Intervention): Participants did not take any preoperative fiber.

INTERVENTIONS:
Dietary Supplement: Psyillium fiber — Participants receive 7 days of psyllium fiber dietary supplement prior to scheduled surgery
  Arms: Intervention - Received fiber

SUMMARY:
Post-operative constipation is one of the most common complaints after pelvic organ prolapse surgery. Psyillum fiber is an FDA-approved, over the counter dietary supplement that is commonly used to treat constipation. The investigators are conducting this study to determine if participants who receive psyllium fiber before surgery have less difficulty with their first bowel movement after surgery.

DETAILED DESCRIPTION:
Post-operative constipation or delay in return to bowel function is a common concern among patients undergoing pelvic reconstructive surgery. A retrospective study reviewing all patient-initiated telephone calls in the postoperative period after pelvic reconstructive surgery found the most frequent concern among patients to be constipation. Moreover, prevention of constipation may help minimize unnecessary pressure and strain on the pelvic floor during post-operative recovery.

There are various strategies for managing post-operative constipation which typically involve medications including stool softeners, laxatives, or stool bulking agents. Several studies have examined the use of these postoperative regimens and have found a shortened time to first bowel movement (BM) with a combination of these medications when compared to placebo.Despite the use of these regimens, most patients do not have their first BM until the second or third postoperative day and this can result in significant distress, discomfort, and fecal impaction.

Postoperative constipation is a multifactorial process and an alternative approach involves consideration of the preoperative period. Preoperative defecation patterns can be a factor in the development of postoperative constipation. We are not aware of any studies looking at the effect of preoperative intervention on postoperative bowel function, particularly the use of preoperative fiber supplementation.

Psyllium fiber is a dietary supplement and stool bulking agent that stimulates peristalsis and improves bowel evacuation. The Western diet is low in fiber and women with pelvic organ prolapse have been found to have lower dietary intake of fiber when compared to controls.8 The primary objective of this study is to evaluate whether the use of preoperative psyllium fiber intake reduces time to first bowel movement after pelvic reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing prolapse repair with or without hysterectomy on the University of Massachusetts urogynecology service

Exclusion Criteria:

* Unable to provide consent
* Under 18 years of age
* Pregnant women
* Prisoners
* As our validated questionnaires are only available in English, we are unable to offer study participation to Non-English speaking subjects
* Because these conditions intrinsically affect bowel function, women with the following will be excluded: history of inflammatory bowel disease, colorectal cancer, rectovaginal fistula, sigmoid resection or rectal surgery
* Because the use of motility agents can affect bowel function and stool transit, women using motility agents such as linaclotide will be excluded.
* Concurrent bowel surgery due to potential effect on the surgical field
* Concurrent anal sphincteroplasty due to potential effect on the surgical field
* Insulin-dependent diabetes mellitus with known gastroparesis as this would affect transit of fiber supplement
* Patients with a history of phenylketonuria as the psyllium fiber supplement we will be using contains phenylalanine
* History of placement of sacral neuromodulating device for indication of fecal incontinence, as this would affect bowel function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Maheshwari, DO, MPH, Principal Investigator — UMass Chan Medical School
Locations (1):
- University of Massachusetts Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramaseshan AS, LaSala C, O'Sullivan DM, Steinberg AC. Patient-Initiated Telephone Calls in the Postoperative Period After Female Pelvic Reconstructive Surgery. Female Pelvic Med Reconstr Surg. 2020 Oct;26(10):626-629. doi: 10.1097/SPV.0000000000000636. PMID 30247168
- [Background] Patel M, Schimpf MO, O'Sullivan DM, LaSala CA. The use of senna with docusate for postoperative constipation after pelvic reconstructive surgery: a randomized, double-blind, placebo-controlled trial. Am J Obstet Gynecol. 2010 May;202(5):479.e1-5. doi: 10.1016/j.ajog.2010.01.003. Epub 2010 Mar 6. PMID 20207340
- [Background] McNanley A, Perevich M, Glantz C, Duecy EE, Flynn MK, Buchsbaum G. Bowel function after minimally invasive urogynecologic surgery: a prospective randomized controlled trial. Female Pelvic Med Reconstr Surg. 2012 Mar-Apr;18(2):82-5. doi: 10.1097/SPV.0b013e3182455529. PMID 22453316
- [Background] Arya LA, Novi JM, Shaunik A, Morgan MA, Bradley CS. Pelvic organ prolapse, constipation, and dietary fiber intake in women: a case-control study. Am J Obstet Gynecol. 2005 May;192(5):1687-91. doi: 10.1016/j.ajog.2004.11.032. PMID 15902178
- [Background] Ballard A, Parker-Autry C, Lin CP, Markland AD, Ellington DR, Richter HE. Postoperative bowel function, symptoms, and habits in women after vaginal reconstructive surgery. Int Urogynecol J. 2015 Jun;26(6):817-21. doi: 10.1007/s00192-015-2634-8. Epub 2015 Feb 12. PMID 25672646
- [Derived] Maheshwari D, Hall CD, Jia X, Tangada A, Wu EK, Leung K, Flynn MK. The Effect of Preoperative Fiber on Postoperative Bowel Function After Pelvic Reconstructive Surgery: A Randomized Controlled Trial. Urogynecology (Phila). 2022 Aug 1;28(8):554-560. doi: 10.1097/SPV.0000000000001203. Epub 2022 May 24. PMID 35649241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention - Received Fiber | Control - Did Not Receive Fiber
Started | 41 | 43
Completed | 35 | 36
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 4 | 4
Not completed — Surgery postponed due to COVID | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention - Received Fiber | Control - Did Not Receive Fiber | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (11.9) | 60 (10.3) | 60.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 33 | 33 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 32 | 31 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
PAC-SYM [Mean (Full Range); unit: units on a scale] — The Patient Assessment of Constipation Symptoms (PAC-SYM) is a validated questionnaire that asks about patient's constipation symptoms. Scores range from 0-48 with lower scores associated with fewer symptoms and higher scores associated with more symptoms
  units on a scale | 0.5 [0.1 to 0.8] | 0.3 [0.2 to 0.7] | 0.3 [0.1 to 0.8]

OUTCOME MEASURES:

1. Primary Outcome: Time to First Bowel Movement After Surgery
Description: Date and time of first bowel movement captured via postoperative bowel diary
Time Frame: Within 7 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Intervention - Received Fiber | Control - Did Not Receive Fiber
Number analyzed (Participants) | 35 | 36
hours | 66.5 (22.7) | 68.3 (25)

2. Secondary Outcome: Pain Associated With First Bowel Movement After Surgery
Description: Pain captured with visual analog scale with 0 being no pain and 10 being worst pain
Time Frame: Within 7 days
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention - Received Fiber | Control - Did Not Receive Fiber
Number analyzed (Participants) | 35 | 36
score on a scale | 2.0 [1.0 to 4.0] | 2.0 [0.0 to 4.0]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Intervention - Received Fiber | Control - Did Not Receive Fiber
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/95/NCT04882995/Prot_SAP_000.pdf